CLINICAL TRIAL: NCT00065715
Title: Placebo: Physician or Pill? A Randomized Trial in a Common Cold Model Funded by NIH NCCAM Under RFA "The Placebo Effect in Clinical Practice"
Brief Title: Echinacea Versus Placebo Effect in Common Cold (Physician Echinacea Placebo)
Acronym: PEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AT001428 (NIH); R01AT001428 (NIH); BarrettB
Record Dates: First submitted 2003-07-31; First posted 2003-08-01 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Common Cold
Keywords: head cold; common cold; echinacea; placebo
MeSH Terms: conditions — Common Cold | interventions — Echinacea extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (No Intervention): No pills
- B (Placebo Comparator): Blinded placebo
  Interventions: Other: Blinded placebo
- C (Experimental): Echinacea - Blinded
  Interventions: Dietary Supplement: Echinacea
- D (Experimental): Echinacea - Unblinded, Open Label
  Interventions: Dietary Supplement: Echinacea

INTERVENTIONS:
Dietary Supplement: Echinacea — Echinacea phytochemical profile Each tablet is comprised of the equivalent of 1275 mg of echinacea root, as follows: A) Echinacea purpurea - 675 mg root yields 112.5 mg dried extract, standardized to contain 2.1mg alkamides. B) Echinacea angustifolia - 600 mg root yields 150 mg dried extract, standardized to contain 2.0 mg alkamides. Each batch of tablets is analyzed by Reversed Phase - High Peformance Liquid Chromatography to determine the levels of alkamides and caffeic derivatives present. Caffeic acid derivative levels are typically as follows: caftaric acid = 0.5 to 2.0 mg/tablet; cichoric acid = 3.4 to 8.5 mg/tablet; chlorogenic acid = < 0.5 mg/tablet; dicaffeoyl quinic acids (including cynarin) = 0.7 to 2.0 mg/tablet; echinacoside = 1.0 to 1.7 mg/tablet
  Arms: C; D
Other: Blinded placebo — Blinded placebo - Coated tablet
  Arms: B

SUMMARY:
The design and interpretation of randomized trials is intimately connected to the use of "placebo". The nature and magnitude of placebo effects, however, is very poorly understood. This study will assess and compare placebo effects and physician interaction effects within a community-acquired common cold model. The goal of this study is to assess two kinds of placebo affects and how physician interaction effects;

1. The effect of receiving blinded placebo, compared to no treatment; and
2. The effect of receiving open-label active Echinacea treatment compared to blinded active treatment.

DETAILED DESCRIPTION:
As per Brief Summary

ELIGIBILITY:
Inclusion criteria:

* Suspected or known cold
* At least one of the following cold symptoms:

nasal discharge, nasal congestion, sneezing, or sore throat

* Enrolled in school, for children 12 to 17 years of age

Exclusion criteria:

* Pregnancy;
* Symptom duration > 36 hrs
* Concurrent use of antibiotics, antivirals, nasal steroids, decongestants or antihistamines;
* Anticipated need for symptom-relieving meds during cold
* Autoimmune/deficiency disease
* History of allergic rhinitis with current eye itching/sneezing
* History of asthma w/current cough/SOB
* Prior study entry
* Allergy to Echinacea

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2003-09; Primary Completion 2008-08 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Duration and severity of illness, as assessed by the Wisconsin Upper Respiratory Symptom Survey (WURSS-21) | twice daily during illness

SECONDARY OUTCOMES:
SF-8 general health-related quality of life | daily during illness
perceived stress PSS-4 | daily during illness
optimism LOT | two days after enrollment
patient satisfaction CARE | after doctor patient interaction
feeling thermometer - EuroQol VAS | daily during illness
IL-8 (inflammatory cytokine)from nasal wash | 2 days after enrollment
neutrophil count from nasal wash | two days after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Barrett, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison Department of Family Medicine, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Montague E, Xu J, Chen PY, Asan O, Barrett BP, Chewning B. Modeling eye gaze patterns in clinician-patient interaction with lag sequential analysis. Hum Factors. 2011 Oct;53(5):502-16. doi: 10.1177/0018720811405986. PMID 22046723
- [Derived] Barrett B, Brown R, Rakel D, Mundt M, Bone K, Barlow S, Ewers T. Echinacea for treating the common cold: a randomized trial. Ann Intern Med. 2010 Dec 21;153(12):769-77. doi: 10.7326/0003-4819-153-12-201012210-00003. PMID 21173411
- See also: Related Info — http://www.fammed.wisc.edu